CLINICAL TRIAL: NCT05893290
Title: How Does Basic Body Awareness Therapy Effect Pain Coping Strategies in Postmenopausal Women? a Randomized Controlled Study
Brief Title: How Does Basic Body Awareness Therapy Effect Pain Coping Strategies in Postmenopausal Women?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Lefke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAYEK022.03
Record Dates: First submitted 2023-05-30; First posted 2023-06-07 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2023-07

CONDITIONS: Low Back Pain; Neck Pain; Menopause
Keywords: Postmenopausal women; Basic body awareness therapy; Pain coping
MeSH Terms: conditions — Low Back Pain; Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Therapeutic Exercise Group (Active Comparator): The therapeutic exercise protocol will be taught to patients in the first session and will be done 3 times a week for 12 weeks.
  Interventions: Other: Therapeutic Exercise Group
- Therapeutic Exercise+Basic Body Awareness (BBAT) Group (Experimental): This group will receive BBAT as well as therapeutic exercises for 3 times a week for 12 week. Therapeutic exercises will include strengthening, stretching, and stabilization exercises. BBAT will include postural alignment, breathing, and cognitive exercises.
  Interventions: Other: Therapeutic Exercise+Basic Body Awareness Therapy Group
- Control Group (No Intervention): This group will not receive any treatment.

INTERVENTIONS:
Other: Therapeutic Exercise Group — Therapeutic exercise sessions will begin with a short educational talk that provides information on proper body mechanics, and the benefits of exercise, followed by simple warm-ups and three different stretching and five different strengthening exercises that emphasize hip, abdominal, and back muscles. The frequency of repetitions of each stretching and strength exercise will be 10 with a holding time of 10 sec. Each set of strengthening exercises will be followed by a different set of stretching exercises. Sessions will end with a short unguided period of deep slow breathing.
  Arms: Therapeutic Exercise Group
Other: Therapeutic Exercise+Basic Body Awareness Therapy Group — This group will receive BBAT as well as therapeutic exercises. Therapeutic exercises will include strengthening, stretching, and stabilization exercises. BBAT will include postural alignment, breathing, and cognitive exercises.
  Arms: Therapeutic Exercise+Basic Body Awareness (BBAT) Group

SUMMARY:
Exercise interventions are deemed essential for the effective management of patients with pain. Various therapy methods have been shown in the literature for pain and coping with pain. However, there is no study investigating the effectiveness of Basic Body Awareness Therapy in pain and coping with pain. In this respect, our study will contribute to the literature. The aim of our study is to compare the effectiveness of Basic Body Awareness Therapy and Therapeutic Exercises on pain coping strategies of Postmenopausal women.

DETAILED DESCRIPTION:
The patients will be randomly assigned into three groups: Therapeutic Exercise (TE) Group, Therapeutic Exercise+Basic Body Awareness (TE+BBAT) Group, and Control Group. Each group will be treated for 12 weeks. Individuals will be evaluated in detail at the beginning and end of the study. The follow-up assessments of the study will be done 3 months after the conclusion of the treatments. Physical and sociodemographic characteristics will be evaluated by dedicated form. The body awareness of the participants will be evaluated Body Awareness Questionnaire (BAQ) developed by Shields, Mallory & Simon in 1989. The pain levels of the PmW will be measured with the Short Form McGill Pain Questionnaire. Pain coping strategies of PmW will be assessed with Pain Coping Inventory (PCI). The Oswestry Low Back Pain Disability Index will be used for evaluating the disability level caused by low back pain. The Neck Disability Index will be used for evaluating the disability level caused by neck pain.

ELIGIBILITY:
Inclusion Criteria: Participants should have;

* Chronic lower back or neck pain lasting at least six months
* Gone through the menopausal transition naturally within the last year
* Not received a physiotherapy approach for pain management in the last six months
* Be able to read and write in Turkish.

Exclusion Criteria:

* Presence of significant neurological disorders
* Presence of serious mental and psychological disorder

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Body Awareness Questionnaire (BAQ) | 3 minutes
  Body awareness of the participants will be evaluated Body Awareness Questionnaire (BAQ) developed by Shields, Mallory & Simon. BAQ is a questionnaire that aims to determine the normal or abnormal sensitivity level of body composition. It consists of four subgroups (Attention to changes in body process and responses, sleep-wake cycle, prediction at onset of illness, prediction of body responses) and a total of 18 statements. The participant will be asked to rate each statement with numbers from one to seven (1 = not at all true for me, 7 = completely true for me). Rating in the survey is done as a total score. It is concluded that the higher the total score to be obtained from the questionnaire, the better the body awareness.
McGill-Short Form Pain Questionnaire | 5 minutes
  The pain levels of the PmW will be measured with the Short Form McGill Pain Questionnaire. The questionnaire, developed by Melzack in 1987 and the validity and reliability of the Turkish version of which was demonstrated in 2007, is widely used in measuring pain. This questionnaire consists of a total of 15 descriptive words to determine the sensory (11 words) and affective (4 words) dimensions of pain. In this section, the severity of pain (0=absent, 1=mild, 2=moderate, 3=severe) is evaluated. In addition, the pain felt at the time of measurement is measured with the Visual Analogue Scale (VAS) and the total pain intensity is measured with a 10-point Likert scale. On this scale, 1 = no pain, 10 = unbearable pain.
Pain Coping Strategies | 5 minutes
  Pain coping strategies of PmW will be assessed with Pain Coping Inventory (PCI). The scale developed by Kraaimaat and Evers evaluates how often chronic pain patients use behavioral and cognitive methods to cope with pain. The original form of the scale includes six dimensions as pain transformation, distraction, reducing demands, retreating, worrying, and resting. Pain transformation, comforting thinking, and distraction are active coping methods; retreat, worrying, and resting are passive coping methods. The scoring options range from 1 (almost none) to 4 (very often).
Oswestry Low Back Pain Disability Index | 5 minutes
  The Oswestry low back pain disability index (OLBPDI), first published in 1980, was developed to assess pain-related disability in people with acute, subacute, or chronic low back pain. It includes 1 item related to pain and 9 items related to activities of daily living (personal care, lifting, walking, sitting, standing, sleeping, social life and travel). Each item is measured on a 6-point ranking scale from best to worst-case scenario. A total score of 0-4 indicates no disability, 5-14 indicates mild disability, 15-24 indicates moderate disability, 25-34 indicates severe functional disability, and 35-50 indicates full functional disability.
Neck Disability Index | 5 minutes
  The questionnaire, which evaluates subjective symptoms and activities of daily living, consists of 10 sections (pain severity, lifting weights, sleep, reading, driving, headache, concentration, work life, personal care, and leisure activities). For each section, there are 6 items ranging from 0-5 points. The total score ranges from 0 to 50 (0: no excuse; 50: maximum excuse). The total score obtained from the questionnaire expresses the severity of neck disability (0-4 points no disability, 5-14 points mild disability, 15-24 points moderate disability, 25-34 points severe disability, and over 35 points total disability).

CONTACTS AND LOCATIONS:
Overall Officials: Beliz Belgen Kaygisiz, PT, PhD, Principal Investigator — European University of Lefke
Locations (1):
- Cyprus Science University, Girne, TRNC, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No